CLINICAL TRIAL: NCT02688101
Title: A Phase 1 Dose-finding and Pharmacokinetic Study of DpC, Administered Orally to Patients With Advanced Solid Tumors
Brief Title: Dose-finding and Pharmacokinetic Study of DpC, Administered Orally to Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Collaborative Medicinal Development Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMD-2015-001
Record Dates: First submitted 2016-01-25; First posted 2016-02-23 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2017-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — di-2-pyridylketone 4-cyclohexyl-4-methyl-3-thiosemicarbazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DpC (Experimental): DpC capsules, administered orally
  Interventions: Drug: DpC

INTERVENTIONS:
Drug: DpC — iron chelator
  Other Names: Dp4cycH4mT

SUMMARY:
Multicenter, open-label, dose-escalation and pharmacokinetic study.

DETAILED DESCRIPTION:
Multicenter, open-label, phase 1 study of DpC administered orally to patients with advanced solid tumors. The study will be conducted in two parts. In the first phase successive cohorts of patients (3+3) will receive escalating doses of DpC until the maximum tolerated dose (MTD) is reached. MTD is based on tolerability observed during the first 28 days of treatment. The second part of the study involves treatment of expansion cohorts (10-15 patients each) in specific indications to confirm the tolerability of treatment at the recommended phase 2 dose and schedule and evaluate evidence of anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study-specific procedures;
* Histologically or cytologically confirmed diagnosis of an advanced or metastatic solid tumor for which standard therapy either does not exist or has proven ineffective, intolerable, or unacceptable for the patient;
* At least one measurable lesion as defined by RECIST v1.1, except for patients with castrate resistant prostate cancer, who may be enrolled with objective evidence of disease per PCWG2 criteria, and patients with ovarian cancer who may be enrolled without measurable disease but who are evaluable by CA125 per GCIC criteria;
* life expectancy at least 3 months;
* ECOG performance status 0-1;
* Adequate bone marrow reserve, cardiac, renal and liver function, defined by
* absolute neutrophil count at least 1.5 x 10(9)/L;
* platelet count at least 100 x 10(9)/L;
* hemoglobin at least 9 g/dL;
* ferritin at least 50 ug/L;
* ECHO shows ejection fraction at least 50% and no evidence of cardiac dysfunction;
* creatinine clearance >50 mL/min (Cockcroft & Gault formula);
* AST/ALT no more than 3 x ULN (5 x ULN if liver or bone involvement);
* serum albumin at least 28 g/L;
* INR no more than 1.5 x ULN;
* At least 3 weeks since chemotherapy, immunotherapy, hormone therapy, r other anticancer therapy or surgical intervention or at least 3 half-lie for monoclonal antibodies;
* Patients with castrate-resistant prostate cancer must maintain ongoing androgen deprivation therapy to provide serum testosterone <50 mg/dL;
* Patients receiving bisphosphonate or denosumab therapy must be on stable doses for at least 4 weeks before initiating study treatment.

Exclusion Criteria:

* Inability to swallow oral medications or presence of a GI disorder deemed to jeopardize intestinal absorption of DpC;
* Persistent grade >1 clinically significant toxicities related to prior anticancer treatment (except alopecia);
* Known primary CNS malignancy or CNS involvement (except for brain mets that have been treated and are stable and patient is off steroids);
* History of prior to concomitant malignancies (other than fully excised non-melanoma skin cancer, cured in situ cervical carcinoma, early stage bladder cancer or DCIS of breast) within 3 years of study entry;
* History of atrial fibrillation or evidence of atrial enlargement on baseline ECHO;
* History of hemoglobinopathy;
* Current use of iron chelation therapy;
* Other serious illness or medial condition;
* Participation in another clinical trial or treatment with any investigational drug within 30 days prior to study entry;
* Current use of anticoagulants at therapeutic levels;
* Pregnant or breast-feeding patients and men and women of child-bearing potential not using effective contraception while on study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose as determined by number of participants at each dose level with dose limiting toxicities | 36 months
  Determine recommended phase 2 dose

SECONDARY OUTCOMES:
Maximum DpC plasma concentration [Cmax] following dosing on Days 1 and 28 based on blood draws taken at 1, 2, 4, 8, and 24 hours after dosing | 30 months
  Maximum DpC plasma concentration
Area under the DpC plasma concentration vs. time curve [AUC] following dosing on Days 1 and 28 based on blood draws taken at 1, 2, 4, 8, and 24 hours after dosing | 30 months
  DpC area under the plasma concentration vs. time curve
Number of patients with tumor responses as assessed by RECIST criteria | 36 months
  number of tumor responses by RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Linda Mileshkin, MD, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (4):
- Australia (4):
  - Lifehouse Cancer Treatment Centre, Sydney, New South Wales
  - Olivia Newton John Cancer Centre, Heidelberg, Victoria
  - Monash Cancer Center, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided